CLINICAL TRIAL: NCT01937819
Title: Patients Judging Dose Adjustment of Bowel Preparation Solution for Bowel Preparation by Using SMARTPHONE Application: A Pilot Study
Brief Title: Patients Judging Bowel Preparation by Using SMARTPHONE Application
Acronym: BPBUSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jongha Park, Study principal investigator, Inje University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SMART-BP01
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: BOWEL PREPARATION (BOWEL CLEANSING)
Keywords: BOWEL PREPARATION; SMARTPHONE APPLICATION

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART arm (Experimental): Using SMARTPHONE application for self judging bowel preparation
  Interventions: Device: SMART arm
- Conventional arm (No Intervention): Non-using SMARTPHONE application for bowel preparation

INTERVENTIONS:
Device: SMART arm — The SMARTPHONE application for self judging bowel preparation by taking the picture of stool form.
  Other Names: SMART-BP
  Arms: SMART arm

SUMMARY:
High-quality bowel preparation is a prerequisite for colonoscopy. Few studies have evaluated visual aids as a means of improving the quality of bowel preparation. We assess the effect of patient-judging dose adjustment of bowel preparation solution for bowel preparation using SMARTPHONE application on the quality of bowel preparation.

DETAILED DESCRIPTION:
This was a randomized, prospective, endoscopist-blinded clinical trial in which the efficacy of SMARTPHONE application on the bowel cleansing was inspected.

A intervention patients take the picture of stool using SMARTPHONE camera application, and then assess the bowel cleansing result. If the result is "Pass", they stop the addition of bowel preparation agent. but the result is "Fail", so they have the additive bowel preparation agent and repeat using the SMARTPHONE application.

After the bowel preparation, Endoscopists, who were blinded to the study group of the patient, immediately completed the Ottawa scale after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are scheduled for colonoscopy Available to use the SMARTPHONE application and smartphone camera

Exclusion Criteria:

* known or suspected bowel obstruction known pregnancy, breast feeding known allergy to PEG presence of severe illness(renal failure, congestive heart failure, liver failure,), refusal of consent to participate in the study not available to use the SMARTPHONE application and SMARTPHONE camera

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
bowel cleaning quality according to Ottawa scale scores | 3 months

SECONDARY OUTCOMES:
The consistency of bowel cleansing result by SMARTPHONE application with Ottawa scale scores by colonoscopy | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Haeundae Paik Hospital, Busan, South Korea